CLINICAL TRIAL: NCT02350933
Title: Endoscopic Evaluation of the Paediatric Airway After Prior Prolonged (>24 h) Tracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Asklepios-Klinik Sankt Augustin (Other); Kinderkrankenhaus Amsterdamer Straße (Unknown); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Endostudy
Record Dates: First submitted 2014-12-12; First posted 2015-01-30 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Intubation; Endoscopy
Keywords: tracheal damages
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0° rigid endoscope (Other): Endoscopy of the trachea is performed using a 0° rigid endoscope
  Interventions: Procedure: Endoscopy

INTERVENTIONS:
Procedure: Endoscopy — A rigid endoscopy of the larynx and the trachea until the carina is performed using a rigid 0° endoscope.

SUMMARY:
The purpose of this study is to determine whether possible damages of the trachea caused by a prior prolonged intubation (> 24h) can be observed by rigid endoscopy of the trachea and if cuffed tracheal tubes cause less damages than cuffed tubes.

DETAILED DESCRIPTION:
The aim of the study is to systematically evaluate airway injury by rigid endoscopy in children (1 month to 16 years of age) with previous prolonged (> 24h) tracheal intubation with a special focus on whether their trachea was intubated with a cuffed or an uncuffed tracheal tube.

After induction of anaesthesia and obtaining venous access, neuromuscular blocking agents are administered and facemask pre-oxygenation occurs for 2 minutes. Direct laryngoscopy is then performed in the preoxygenated, paralysed and conventionally monitored patient to obtain a direct vision. Then a rigid endoscope with endoscopy camera is carefully guided through the larynx down to the carina and drawn back under monitor vision with electronic recording.

An International Study Board Committee (assessor board) will assess the endoscopic records in a blinded manner using a systematic grading system.

Beside tracheal tube type, factors such as intubator, sedation management, age, length of intubation, nasal or oral intubation and time point of endoscopy will affect presence, absence or incidence of potential airway injuries caused by prolonged tracheal intubation. Thus it is difficult to perform a power calculation to figure out number of patients to demonstrate or exclude a statistically significant difference between tube types. Using the incidence of subglottic stenosis, as the worst case scenario outcome after longterm intubation, an incidence of less than 2 % seems to be reasonable in uncuffed tracheal tubes.So the primary hypothesis to be tested is equivalence in major complication rates defined as subglottic stenosis comparing cuffed versus uncuffed tracheal tubes.

Specifically, the primary hypothesis relates to the main outcome criteria of this study, which is subglottic stenosis after longterm intubation. The null-hypothesis Ho is defined as no difference in the incidence rates of subglottic stenosis between cuffed and uncuffed groups. The null-hypothesis (Ho: μ-Diff = 0) will be compared with the alternative hypothesis (H1: μ-Diff <> 0). The study is designed to detect a clinically unacceptable deterioration of 4% above the baseline airway-injury rate of 2% when using uncuffed tubes with a power of 80% and a type I error probability of less than 5%. Sample sizes of 376 from the cuffed group and 376 from the uncuffed group achieve 80% power at a 5% significance level using a one-sided equivalence test of proportions when the proportion in the standard group (uncuffed TT) is 0.02 and the proportion in the experimental group (cuffed TT) being tested for equivalence is 0.02 and the maximum allowable increase between these proportions that still results in equivalence (the range of equivalence) is 0.04. In total 1000 patients with prior long-term intubation (> 24 hours) using a cuffed (500) or an uncuffed (500) tracheal tube will be recruited / included from different study centres.

ELIGIBILITY:
Inclusion Criteria:

* Planned elective intervention/surgery/diagnostics/endoscopy and general anaesthesia with airway instrumentation involving muscle paralysis in children, aged 1 month (UK) or from birth (other centers) to 16 years having prior prolonged (≥ 24h) tracheal intubation (s) during ICU-stay (s) within the study centre (patients for diagnosis/treatment of stridor are also included (see exclusion criteria also below)).
* No known risk for regurgitation
* Written parental consent
* American Society of Anesthesiologists (ASA) physical status < IV

Exclusion Criteria:

* No parental written consent
* Known airway anomalies associated with syndromes
* Known or suspected difficult intubation
* Emergency surgery or intervention
* Full stomach and/or at risk for regurgitation
* ASA physical status IV and higher
* Patients with current or prior tracheostomy
* Known, suspected or potential cervical spine pathology (e.g. Down's Syndrome)
* Insufficient clinical details from previous prolonged intubation

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with evidence of subglottic stenosis after longterm intubation with cuffed versus uncuffed tracheal tubes | After an average induction period of 10 min of an anesthesia with a planned intubation after the endoscopy
  An International Study Board Committee (assessor board) will assess the endoscopic records in a blinded manner using a systematic grading system.

SECONDARY OUTCOMES:
Numbers of prior intubations | Retrospective data analysis of former intubations is performed within two years after the endoscopy
  Numbers of shortterm and prolonged (>24h) and numbers of intubations with cuffed and uncuffed tubes are listed
Duration of prior longterm intubation | Retrospective data analysis of former intubations is performed within two years after the endoscopy
Reason for prior longterm intubation | Retrospective data analysis of former intubations is performed within two years after the endoscopy
  Reason for prior longterm intubation is look up in patient's medical records.
Route of prior longterm intubation | Retrospective data analysis of former intubations is performed within two years after the endoscopy
  Route of prior longterm intubation (nasal or oral) is look up in patient's medical records.
Tube type used for prior longterm intubation | Retrospective data analysis of former intubations is performed within two years after the endoscopy
  Tube type used for prior longterm intubation (cuffed or uncuffed) is look up in patient's medical records.
Tube brand used for prior longterm intubation | Retrospective data analysis of former intubations is performed within two years after the endoscopy
  Tube brand used for prior longterm intubation is look up in patient's medical records.
Tube size used for prior longterm intubation | Retrospective data analysis of former intubations is performed within two years after the endoscopy
  Tube size (inner diameter) used for prior longterm intubation is look up in patient's medical records.
Site of prior longterm intubation | Retrospective data analysis of former intubations is performed within two years after the endoscopy
  Site of prior longterm intubation is look up in patient's medical records.
Maximal cuff pressure during prior longterm intubation | Retrospective data analysis of former intubations is performed within two years after the endoscopy
  Maximal cuff pressure in cmH2O during longterm intubation is look up in patient's medical records.
Number of patients with a stridor event after extubation of prior longterm intubation | Retrospective data analysis of former intubations is performed within two years after the endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Markus Weiss, Prof., Principal Investigator — University Children's Hospital, Zurich
Locations (5):
- Germany (2):
  - Kinderkrankenhaus Amsterdamer Straße, Cologne, North Rhine-Westphalia
  - Asklepios Kinderklinik Sankt Augustin, Sankt Augustin, North Rhine-Westphalia
- Erasmus Medical Center, Sophia Children's Hospital, Rotterdam, Netherlands
- University Children's Hospital, Zurich, Switzerland
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, United Kingdom